CLINICAL TRIAL: NCT01682720
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of GS-7977+Ribavirin for 12 Weeks in Treatment Naive and Treatment Experienced Subjects With Chronic Genotype 2 or 3 HCV Infection.
Brief Title: Sofosbuvir and Ribavirin in Treatment-Naive and Treatment-Experienced Subjects With Chronic Genotype 2 or 3 HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-334-0133; 2012-001942-16 (EudraCT Number)
Record Dates: First submitted 2012-09-05; First posted 2012-09-11 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Hepatitis C
Keywords: HCV; Genotype 2; Genotype 3
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo 12 Weeks (GT2/3) (Placebo Comparator): Placebo to match SOF + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks in participants with genotype 2 or 3 HCV infection.
  Interventions: Drug: Placebo to match SOF; Drug: Placebo to match RBV
- SOF 12 Weeks (GT2/3) (Experimental): Placebo to match SOF + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks in participants with genotype 2 or 3 HCV infection.
  Interventions: Drug: SOF; Drug: RBV
- SOF 24 Weeks (GT3) (Experimental): SOF 400 mg tablet once daily + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 24 weeks in participants with genotype 3 HCV infection.
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: SOF 12 Weeks (GT2/3); SOF 24 Weeks (GT3)
Drug: RBV — Ribavirin (RBV) 200 mg tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: SOF 12 Weeks (GT2/3); SOF 24 Weeks (GT3)
Drug: Placebo to match SOF — Placebo to match SOF administered orally once daily
  Arms: Placebo 12 Weeks (GT2/3)
Drug: Placebo to match RBV — Placebo to match RBV administered orally in a divided daily dose
  Arms: Placebo 12 Weeks (GT2/3)

SUMMARY:
This study will evaluate the safety, tolerability, and antiviral efficacy of GS-7977 with ribavirin (RBV) in participants with genotype 2 or 3 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 with chronic genotype 2 or 3 HCV infection
* HCV RNA > 10,000 IU/mL at screening
* Subjects must be treatment naive or treatment experienced
* Presence or absence of cirrhosis; a liver biopsy may be required
* Healthy according to medical history and physical examination with the exception of HCV diagnosis
* Agree to use two forms of highly effective contraception for the duration of the study and 6 months after the last dose of study medication

Exclusion Criteria:

* Prior use of any other inhibitor of the HCV NS5B Polymerase
* History of any other clinically significant chronic liver disease
* Evidence of or history of decompensated liver disease
* HIV or chronic hepatitis B virus (HBV) infection
* Hepatocellular carcinoma (HCC) or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of immunosuppressive agents or immunomodulatory agents
* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study or not be in the best interest of the subject in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Hyland, DPhil, Study Director — Gilead Sciences Study Director
Locations (77):
- Austria (3):
  - Medizinische Universitat Graz, Graz
  - Medizinische Universitat Wien, Vienna
  - Wilhelminenspital, Vienna
- Estonia (2):
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- France (15):
  - CHRU de Lille, Hopital Claude Huriez, CHRU Lille
  - CHU Estaing, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Henri Mondor, Créteil
  - Département Hépatogastroentérologie - CHU de Grenoble, Grenoble
  - Hopital Saint Joseph, Marseille
  - Hopital Saint Eloi, Montpellier
  - Hopital de l Archet 2, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Pitie Salpetriere, Paris
  - Hopitaux Universitaires, Paris
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - USN, Pessac
  - CHU Pontchaillou - Hématologie Clinique, Rennes
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - CHU de Nancy, Hôpital de Brabois, Vandœuvre-lès-Nancy
- Germany (14):
  - Praxiszentrum, Freiburg im Breisgau, Baden-Wurttemberg
  - Leber- and Studienzentrum am Checkpoint, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Heinrich Heine Unversitat, Düsseldorf
  - JWG-Universität Frankfurt, Frankfurt am Main
  - Asklepios Klinik Sankt Georg H, Hamburg
  - Universitatsklinikum, Hamburg
  - Medizinische Hochschule Hannov, Hanover
  - Medizinische Klinik IV, Dep. o, Heidelberg
  - Gastroenterologische Gemeinsch, Herne
  - Leberstudienzentrum Kiel, Kiel
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Universität Münch, München
  - Centrum fuer interdisziplinaere Medizin Muenster GmbH, Münster
- Italy (12):
  - Ospedale Casa Sollievo, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera di Bologna - Policlinico S. Orsola Malpighi, Bologna
  - Ospedale S. Annunziata, Florence
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Fondazione IRCCS CA Granada - Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Ospedale Niguarda Cà Granda, Milan
  - University of Padova, Padua
  - University of Palermo, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione PTV - Policlinico Tor Vergata, Roma
  - INMI "Lazzaro Spallanzani" I.R.C.C.S., Roma
  - Azienda Ospedaliera Universitaria San Giovanni Battista di Torino, Torino
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - UMC St. Radboud - Gastroenterology, Nijmegen
  - Erasmus MC, Rotterdam
- Poland (4):
  - Wojewodzki Szpital Specjalistyczny im Dluskeigo, Bialystok
  - Wojewodzki Specjalistyczny Szpital im. W. Bieganskiego, Lodz
  - SP ZOZ Wojewodzki Szpital Zakazny w Warszawie, Warsaw
  - NZOZ Centrum Badan Klinicznych, Wroclaw
- Spain (9):
  - Hospital Universitari Vall d'H, Barcelona
  - Hospital Casa de la Maternidad, Barcelona
  - Hospital Carlos III, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Puerta de Hierro Maja, Majadahonda
  - Complejo Hospitalario de Especialidades Virgen de la Victoria, Málaga
  - Hospital Universitario Marques, Santander
  - Valme Hospital, Seville
  - Hospital General Universitario de Valencia, Valencia
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skånes Universitetssjukhus, Lund, Lund
  - Skanes Universitetssjukhus, Malmo
  - Karolinska Instituet, Stockholm
- United Kingdom (10):
  - University of Birmingham, Edgbaston, Birmingham
  - Southampton University Hospital NHS Trust, Southhampton, Hampshire
  - King's College Hospital, Denmark Hill, London
  - The Liver Unit, Paddington, London
  - North Manchester General Hospital, Crumpsall, Manchester
  - Bristol Royal Infirmary, Bristol
  - Queen Marys University of London, London
  - Royal Free Hospital and University College London Hospital, London
  - Chelsea & Westminster Hospital, London
  - Nottingham University Hospitals-NHS, Nottingham

REFERENCES:
- [Result] Zeuzem S, Dusheiko GM, Salupere R, Mangia A, Flisiak R, Hyland RH, Illeperuma A, Svarovskaia E, Brainard DM, Symonds WT, Subramanian GM, McHutchison JG, Weiland O, Reesink HW, Ferenci P, Hezode C, Esteban R; VALENCE Investigators. Sofosbuvir and ribavirin in HCV genotypes 2 and 3. N Engl J Med. 2014 May 22;370(21):1993-2001. doi: 10.1056/NEJMoa1316145. Epub 2014 May 4. PMID 24795201
- [Derived] Younossi ZM, Stepanova M, Sulkowski M, Naggie S, Puoti M, Orkin C, Hunt SL. Sofosbuvir and Ribavirin for Treatment of Chronic Hepatitis C in Patients Coinfected With Hepatitis C Virus and HIV: The Impact on Patient-Reported Outcomes. J Infect Dis. 2015 Aug 1;212(3):367-77. doi: 10.1093/infdis/jiv005. Epub 2015 Jan 12. PMID 25583164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 77 study sites in Europe. The first participant was screened on 19 September 2012. The last participant observation occurred on 08 January 2014.
Pre-assignment Details: * 475 participants were screened and 421 were randomized.
  * 419 participants were randomized and received at least 1 dose of study drug (Safety Analysis Set).
  * 334 participants with genotype 2 or 3 hepatitis C virus (HCV) infection were randomized and received at least 1 dose of sofosbuvir (Full Analysis Set).
Groups:
- Placebo 12 Weeks (GT2/3): Placebo to match sofosbuvir (SOF) + placebo to match ribavirin (RBV) for 12 weeks in participants with genotype (GT)2 or 3 HCV infection.
- SOF 12 Weeks (GT2): SOF 400 mg tablet once daily + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks in participants with genotype 2 HCV infection.
- SOF 12 Weeks (GT3): SOF 400 mg tablet once daily + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks in participants with genotype 3 HCV infection.
Period: Overall Study
Arm/Group | Placebo 12 Weeks (GT2/3) | SOF 12 Weeks (GT2) | SOF 12 Weeks (GT3) | SOF 24 Weeks (GT3)
Started | 85 | 74 | 12 | 250
Included in Full Analysis Set | 0 | 73 | 11 | 250
Completed | 0 | 69 | 5 | 211
Not Completed | 85 | 5 | 7 | 39
Not completed — Randomized but Not Treated | 0 | 1 | 1 | 0
Not completed — Terminated by Sponsor | 83 | 0 | 0 | 0
Not completed — Efficacy Failure | 0 | 3 | 3 | 30
Not completed — Lost to Follow-up | 1 | 1 | 0 | 6
Not completed — Subject Withdrew Consent | 0 | 0 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Groups:
- Placebo 12 Weeks (GT2/3): Placebo to match SOF + placebo to match RBV for 12 weeks in participants with genotype 2 or 3 HCV infection.
- Total: Total of all reporting groups
Arm/Group | Placebo 12 Weeks (GT2/3) | SOF 12 Weeks (GT2) | SOF 12 Weeks (GT3) | SOF 24 Weeks (GT3) | Total
Number analyzed (Participants) | 85 | 73 | 11 | 250 | 419
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10.5) | 58 (10.1) | 46 (8.8) | 48 (10.1) | 50 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 5 | 95 | 169
  Male | 49 | 40 | 6 | 155 | 250
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 10 | 6 | 1 | 36 | 53
  Not Hispanic or Latino | 71 | 65 | 10 | 203 | 349
  Not Permitted | 4 | 2 | 0 | 11 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 5 | 0 | 0 | 6
  White | 81 | 65 | 11 | 236 | 393
  Asian | 3 | 1 | 0 | 9 | 13
  Not permitted | 0 | 2 | 0 | 5 | 7
Region of Enrollment [Number; unit: participants]
  France | 13 | 15 | 0 | 53 | 81
  Estonia | 3 | 2 | 4 | 6 | 15
  Spain | 11 | 5 | 1 | 31 | 48
  Poland | 4 | 0 | 0 | 18 | 22
  Austria | 4 | 2 | 0 | 12 | 18
  Netherlands | 5 | 6 | 0 | 14 | 25
  Germany | 14 | 8 | 1 | 46 | 69
  United Kingdom | 17 | 3 | 4 | 31 | 55
  Italy | 9 | 25 | 1 | 27 | 62
  Sweden | 5 | 7 | 0 | 12 | 24
HCV Genotype [Number; unit: participants]
  Genotype 2 | 18 | 73 | 0 | 0 | 91
  Genotype 3 | 67 | 0 | 11 | 250 | 328
Liver Cirrhosis [Number; unit: participants]
  No | 68 | 62 | 9 | 190 | 329
  Yes | 17 | 11 | 2 | 60 | 90
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 22 | 24 | 4 | 86 | 136
    CT | 49 | 41 | 4 | 131 | 225
    TT | 14 | 8 | 3 | 33 | 58
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.69) | 6.5 (0.70) | 6.2 (0.77) | 6.3 (0.74) | 6.4 (0.72)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 21 | 16 | 4 | 72 | 113
  ≥ 6 log10 IU/mL | 64 | 57 | 7 | 178 | 306
Prior HCV Treatment Experience [Number; unit: participants]
  Experienced | 50 | 41 | 9 | 145 | 245
  Naive | 35 | 32 | 2 | 105 | 174
Response to prior HCV treatment [Number; unit: participants] — Only participants who were treatment-experienced at baseline were analyzed.
  participants
    Interferon intolerant | 0 | 3 | 0 | 10 | 13
    Nonresponse | 18 | 10 | 4 | 41 | 73
    Relapse/Breakthrough | 32 | 28 | 5 | 94 | 159
Interferon Eligibility [Number; unit: participants] — Only participants who were treatment-naive at baseline were analyzed.
  participants
    Interferon eligible | 30 | 27 | 2 | 94 | 153
    Interferon ineligible | 5 | 5 | 0 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ, ie, < 25 IU/mL) 12 weeks following the last dose of study drug. Data for this outcome measure was not collected for the Placebo 12 Weeks (GT2/3) group.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants with genotype 2 or 3 HCV infection were randomized and received at least 1 dose of SOF.
Measure: Number; unit: percentage of participants
Arm/Group | SOF 12 Weeks (GT2) | SOF 12 Weeks (GT3) | SOF 24 Weeks (GT3)
Number analyzed (Participants) | 73 | 11 | 250
percentage of participants | 93.2 | 27.3 | 85.2

2. Primary Outcome: Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The percentage of participants experiencing an adverse event leading to permanent discontinuation of study drug(s) was analyzed.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- SOF 12 Weeks (GT2/3): SOF 400 mg tablet once daily + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks in participants with genotype 2 or 3 HCV infection.
Arm/Group | Placebo 12 Weeks (GT2/3) | SOF 12 Weeks (GT2/3) | SOF 24 Weeks (GT3)
Number analyzed (Participants) | 85 | 84 | 250
percentage of participants | 1.2 | 1.2 | 0.4

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 was defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively. Data for this outcome measure was not collected for the Placebo 12 Weeks (GT2/3) group.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set: participants with genotype 2 or 3 HCV infection were randomized and received at least 1 dose of SOF.
Measure: Number; unit: percentage of participants
Arm/Group | SOF 12 Weeks (GT2) | SOF 12 Weeks (GT3) | SOF 24 Weeks (GT3)
Number analyzed (Participants) | 73 | 11 | 250
percentage of participants
  SVR4 | 93.2 | 45.5 | 87.2
  SVR24 | 93.2 | 27.3 | 84.4

4. Secondary Outcome: Percentage of Participants Experiencing Viral Breakthrough or Viral Relapse
Description: Viral breakthrough was defined as having confirmed detectable HCV RNA levels (HCV RNA > LLOQ) after having previously had undetectable HCV RNA levels (HCV RNA < LLOQ) while on treatment.
  Viral relapse was defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) at end of treatment, but did not achieve an SVR.
  Data for this outcome measure was not collected for the Placebo 12 Weeks (GT2/3) group.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set: participants with genotype 2 or 3 HCV infection were randomized and received at least 1 dose of SOF.
Measure: Number; unit: percentage of participants
Arm/Group | SOF 12 Weeks (GT2) | SOF 12 Weeks (GT3) | SOF 24 Weeks (GT3)
Number analyzed (Participants) | 73 | 11 | 250
percentage of participants
  Viral breakthrough | 0 | 0 | 0.4
  Viral relapse | 6.8 | 54.5 | 14.0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24 plus 30 days
Description: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug.
Arm/Group | Placebo 12 Weeks (GT2/3) | SOF 12 Weeks (GT2/3) | SOF 24 Weeks (GT3)
Serious Adverse Events (participants affected / at risk) | 2/85 | 0/84 | 10/250
Other Adverse Events (participants affected / at risk) | 60/85 | 72/84 | 229/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 12 Weeks (GT2/3) (N=85) | SOF 12 Weeks (GT2/3) (N=84) | SOF 24 Weeks (GT3) (N=250)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Adenocarcinoma of colon (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Complex regional pain syndrome (Nervous system disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 12 Weeks (GT2/3) (N=85) | SOF 12 Weeks (GT2/3) (N=84) | SOF 24 Weeks (GT3) (N=250)
Anaemia (Blood and lymphatic system disorders) | 1 | 6 | 17
Nausea (Gastrointestinal disorders) | 9 | 26 | 33
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 30
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7 | 15
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 21
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 15
Constipation (Gastrointestinal disorders) | 1 | 2 | 13
Fatigue (General disorders) | 16 | 19 | 75
Asthenia (General disorders) | 4 | 21 | 53
Irritability (General disorders) | 3 | 4 | 26
Influenza like illness (General disorders) | 5 | 1 | 16
Pyrexia (General disorders) | 2 | 7 | 9
Chest pain (General disorders) | 0 | 5 | 5
Nasopharyngitis (Infections and infestations) | 9 | 4 | 36
Influenza (Infections and infestations) | 0 | 6 | 12
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 13
Headache (Nervous system disorders) | 23 | 24 | 74
Dizziness (Nervous system disorders) | 2 | 5 | 19
Disturbance in attention (Nervous system disorders) | 2 | 1 | 15
Insomnia (Psychiatric disorders) | 2 | 9 | 41
Sleep disorder (Psychiatric disorders) | 4 | 4 | 23
Anxiety (Psychiatric disorders) | 2 | 1 | 13
Depressed mood (Psychiatric disorders) | 2 | 1 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 12 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 27
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 20 | 67
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 8 | 31
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 24
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years